CLINICAL TRIAL: NCT00356460
Title: A Phase 1 Study of the Safety and Efficacy of GC1008: A Human Anti Transforming Growth Factor-beta (TGFβ) Monoclonal Antibody in Patients With Advanced Renal Cell Carcinoma or Malignant Melanoma
Brief Title: Safety and Efficacy Study of GC1008 to Treat Renal Cell Carcinoma or Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC100800305; NCT00381745 (obsolete NCT alias)
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Carcinoma, Renal Cell; Melanoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma | interventions — Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 - Part 1 (Experimental): Dose Group
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody
- 2 - Part 1 (Experimental): Dose Group
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody
- 3 - Part 1 (Experimental): Dose Group
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody
- 4 - Part 1 (Experimental): Dose Group
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody
- 5 - Part 1 (Experimental): Dose Group
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody
- 6 - Part 1 (Experimental): Dose Group
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody
- 1 (Part 2) (Experimental)
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ ) Monoclonal Antibody
- 2 (part 2) (Experimental)
  Interventions: Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody

INTERVENTIONS:
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 0.1 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 0.1 mg/kg IV (one dose every 14 days)
  Arms: 1 - Part 1
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 0.3 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 0.3 mg/kg IV (one dose every 14 days)
  Arms: 2 - Part 1
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 1.0 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 1.0 mg/kg IV (one dose every 14 days)
  Arms: 3 - Part 1
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 3.0 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 3.0 mg/kg IV (one dose every 14 days)
  Arms: 4 - Part 1
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 10.0 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 10.0 mg/kg IV (one dose every 14 days)
  Arms: 5 - Part 1
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 15.0 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 15.0 mg/kg IV (one dose every 14 days)
  Arms: 6 - Part 1
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ ) Monoclonal Antibody — 1 dose of 15.0 mg/kg IV followed by a 28 day observation period and then 3 additional doses of 15.0 mg/kg IV (one dose every 14 days)
  Arms: 1 (Part 2)
Biological: GC1008 Human Anti Transforming Growth Factor _Beta (TGFβ) Monoclonal Antibody — 1 dose of 15.0 or 10.0 mg/kg IV (based on safety profile of part 2, cohort 1) followed by a 28 day observation period and then 3 additional doses of 15.0 or 10.0 mg/kg IV (one dose every 14 days)
  Arms: 2 (part 2)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of GC1008, a human anti-transforming growth factor-beta (TGFβ) monoclonal antibody in previously treated patients with locally advanced or metastatic renal cell carcinoma or malignant melanoma.

DETAILED DESCRIPTION:
Transforming growth factor-beta (TGFβ) is a cytokine which is often over-expressed and over-produced by malignancies and has been implicated as an important factor in promoting the growth, progression, and metastatic potential of advanced cancers. In preclinical studies, TGFβ can act to promote tumor cell migration/invasiveness, influence tumor stroma (by increasing extracellular matrix production, cytokine secretion, and angiogenesis), and suppress anti-tumor immunity. The purpose of this study is to investigate the clinical use of GC1008, a human monoclonal antibody capable of binding and neutralizing all isoforms of TGFβ.

This is a Phase 1 multi-center, open-label, dose-escalation study designed to characterize the safety, tolerability, pharmacokinetic, pharmacodynamic, and potential anti-tumor activity of GC1008, in patients with histologically confirmed, locally advanced and surgically inoperable or metastatic renal cell carcinoma (RCC) or malignant melanoma. Patients with RCC must have failed at least 1 prior therapy and patients with renal cell carcinoma must have failed either sorafenib or sunitinib. Other qualifying prior therapies includes any medical, surgical, radiation or investigational approaches used for potential therapeutic benefit (but not for diagnostic purposes) in patients with advanced disease. Patients may receive up to 4 intravenous infusions of GC1008, and patients with stable disease, with an objective tumor response or with clinical benefit may be eligible to receive extended therapy. For part 2 of the study, only patients with malignant melanoma will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* In Part 1, Dose Escalation: Patients with histologically confirmed, locally advanced & surgically inoperable or metastatic renal cell carcinoma or malignant melanoma are eligible.
* In Part 2, Patient Expansion: Patients with histologically confirmed, locally advanced and surgically inoperable or metastatic malignant melanoma are eligible.
* In both part 1 and 2: All patients must have failed ≥ 1 prior therapy and potential patients may not be eligible for curative intent treatment (e.g., potentially curative surgical resection or chemotherapy). Other qualifying therapies include any medical, surgical, radiation, or investigational approach used for potential therapeutic benefit (but not for diagnostic purposes) in patients with advanced disease.In addition, In Part 1, Patients with renal cell carcinoma must have failed temsirolimus and either sorafenib or sunitinib as part of their prior therapies.
* Expected survival ≥5 months
* Eastern cooperative oncology Group (ECOG) Performance Status 0 to 2.
* Measurable disease as defined by RECIST
* Laboratory: a. Serum albumin > or = 3.0 g/dL. b. Marrow: Hemoglobin > or =10.0 g/dL, absolute neutrophil count (ANC) > or = 1,500/mm3, and platelets > or = 100,000/mm3. c. Hepatic: Serum total bilirubin < or = 1.5 x upper limit of normal (ULN) (Patients with Gilbert's Disease may be included if their total bilirubin is < or = 3.0 mg/dL.), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) < or = 2.5 x ULN. If the patient has known liver metastases, an ALT and/or AST < or =5 x ULN are allowed. d. Renal: If negative proteinuria on urine dipstick, serum creatinine (sCr) < 2 mg/dL or urine creatinine clearance > or = 60 mL/min. If urine is 1+ positive (30 mg/dL), urine protein must be < or =1 g/24 hours and measured creatinine clearance > or = 60 mL/min. e. Prothrombin time (PT) and partial thromboplastin time (PTT) within normal ranges. f. Negative tests (antibody and/or antigen) for hepatitis viruses B and C and HIV
* At the time of enrollment, patients must be >4 wks since major surgery, radiotherapy, chemotherapy (> or =6 wks if they were treated with a nitrosourea, mitomycin, or monoclonal antibodies such as bevacizumab), immunotherapy, or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to< or = Grade 1, exclusive of alopecia. Concurrent cancer therapy is not permitted. (In patients who received long acting agents, a treatment-free interval of 2 half-lives should be considered.)
* Patients must be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney.
* Male and female patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the experimental drug, and for at least 3 months after the last treatment. Female patients of child-producing potential must have a negative serum pregnancy test confirmed within 7 days of receiving the initial dose of GC1008 therapy.
* Documentation of flu vaccination if enrolled during flu season (as defined by the availability of vaccine). Otherwise, patient should receive the current flu vaccine > or = 1 wk before beginning GC1008 therapy.
* Pre-treatment tumor samples, such as paraffin blocks or unstained slides, must be available for analyses.

Exclusion Criteria:

* Central nervous system (CNS) metastases, meningeal carcinomatosis, malignant seizures, or a disease that either causes or threatens neurologic compromise (e.g., unstable vertebral metastases).
* History of ascites or pleural effusions, unless successfully treated, completely resolved, and the patient has not been treated for these conditions for >4 months.
* Active thrombophlebitis, thromboembolism, hypercoagulability states, bleeding, or use of anti-coagulation therapy (including anti-platelet agents). Patients with a history of deep venous thrombosis may participate if successfully treated, completely resolved, and no treatment has been given for >4 months.
* Hypercalcemia: Calcium >11.0 mg/dL (2.75 mmol/L) unresponsive or uncontrolled in response to standard therapy (e.g., bisphosphonates).
* Pregnant or nursing women, due to the unknown effects of GC1008 on the developing fetus or newborn infant.
* Patients diagnosed with another malignancy - unless following curative intent therapy, the patient has been disease free for at least 5 yrs and the probability of recurrence of the prior malignancy is <5%. Patients with curatively treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are eligible for this study.
* Patients with an organ transplant, including those that have received an allogeneic bone marrow transplant.
* Use of investigational agents within 4 wks prior to study enrollment (within 6 wks if the treatment was with a long-acting agent such as a monoclonal antibody).
* Patients on immunosuppressive therapy including: a. Systemic corticosteroid therapy for any reason, including replacement therapy for hypoadrenalism, pAtients receiving inhaled or topical corticosteroids may participate. b. Patients receiving cyclosporine A, tacrolimus, or sirolimus are not eligible for this study.
* Significant or uncontrolled medical illness, such as congestive heart failure (CHF), myocardial infarction, symptomatic coronary artery disease, significant ventricular arrhythmias within the last 6 months, or significant pulmonary dysfunction. Patients with a remote history of asthma or active mild asthma may participate.
* Active infection, including unexplained fever (temperature >38.1 degrees C) or antibiotic therapy within 1 wk prior to enrollment.
* Systemic autoimmune disease (e.g., systemic lupus erythematosus, active rheumatoid arthritis, etc.).
* A known allergy to any component of GC1008.
* Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion. Examples of significant problems include, but are not limited to: a. Other serious non-malignancy-associated medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis) or significantly increase the risk of SAEs. b. Any condition psychiatric or otherwise, that would preclude informed consent, consistent follow-up, or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment). c. Patients currently abusing drugs or alcohol or, in the opinion of the investigator, at high risk for poor compliance.
* Part 2 only: Prior therapy with a TGFB antagonist, such as an antibody, receptor, or kinase inhibitor or anti-sense therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Part 1: To assess the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and safety of GC1008 in patients with locally advanced or metastatic renal cell carcinoma or malignant melanoma. | up to 2.5 years
Part 1: To assess dose-limiting toxicity of GC1008 in patients with locally advanced metastatic renal cell carcinoma or malignant melanoma. | up to 2.5 years
Part 1: To assess the safety of GC1008 in patients with locally advanced or metastatic renal cell carcinoma or malignant melanoma. | up to 2.5
Part 2: To assess the safety of GC1008 following multiple doses at 15 mg/kg (or 10 mg/kg depending on the safety review of the first cohort of 6 patients at 15 mg/kg) in patients with locally advanced or metastatic malignant melanoma. | Up to 2 years

SECONDARY OUTCOMES:
Part 1 & 2: To assess possible surrogate markers that might predict clinical efficacy by obtaining skin (part 2), tumor and blood samples for exploratory biomarker analyses. | up to 2.5 years
Part 1 & 2: To obtain pharmacokinetic (PK) and pharmacodynamic (PD) data on GC1008. | up to 2.5 years
Part 1 & 2: To evaluate tumor response as a preliminary assessment of clinical activity. | up to 2.5 years
Part 2: To evaluate the relationship between GC1008 exposure, clinical response, and the development of skin lesions. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (6):
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Dana Farber/Harvard Cancer Center, Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Cambridge, Massachusetts
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Morris JC, Tan AR, Olencki TE, Shapiro GI, Dezube BJ, Reiss M, Hsu FJ, Berzofsky JA, Lawrence DP. Phase I study of GC1008 (fresolimumab): a human anti-transforming growth factor-beta (TGFbeta) monoclonal antibody in patients with advanced malignant melanoma or renal cell carcinoma. PLoS One. 2014 Mar 11;9(3):e90353. doi: 10.1371/journal.pone.0090353. eCollection 2014. PMID 24618589
- [Derived] Berzofsky JA, Wood LV, Terabe M. Cancer vaccines: 21st century approaches to harnessing an ancient modality to fight cancer. Expert Rev Vaccines. 2013 Oct;12(10):1115-8. doi: 10.1586/14760584.2013.836906. No abstract available. PMID 24124874